CLINICAL TRIAL: NCT04543877
Title: WHNRC (Western Human Nutrition Research Center) Fiber Intervention Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: FL113
Record Dates: First submitted 2020-08-24; First posted 2020-09-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Inflammation; Vaccine; Intestinal Permeability; Typhoid Fever
Keywords: Gastrointestinal Health; Intestinal Permeability; Vaccine Response; Inflammation; Ty21a Typhoid Vaccine; Typhoid Fever; Microbiome; Bifidobacterium
MeSH Terms: conditions — Inflammation; Typhoid Fever | interventions — Inulin; maltodextrin; Ty21a typhoid vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inulin and Ty21a Vaccine (Experimental): Participants will consume 12 grams/day of inulin for 3 weeks before the administration of the Ty21a vaccine, 1 week during the vaccine, and 1 week after the vaccine for a total of 5 weeks.
  Interventions: Dietary Supplement: Inulin; Biological: Ty21a Typhoid Fever Vaccine
- Maltodextrin and Ty21a Vaccine (Placebo Comparator): Participants will consume 12 grams/day of maltodextrin (control) for 3 weeks before the administration of the Ty21a vaccine, 1 week during the vaccine, and 1 week after the vaccine for a total of 5 weeks.
  Interventions: Dietary Supplement: Maltodextrin; Biological: Ty21a Typhoid Fever Vaccine

INTERVENTIONS:
Dietary Supplement: Inulin — Consume 12 grams/day of inulin for 5 weeks (Day 9 - 43).
  Other Names: Orafti GR
  Arms: Inulin and Ty21a Vaccine
Dietary Supplement: Maltodextrin — Consume 12 grams/day of maltodextrin for 5 weeks (Day 9 - 43).
  Other Names: Maltrin M100
  Arms: Maltodextrin and Ty21a Vaccine
Biological: Ty21a Typhoid Fever Vaccine — All participants will receive the vaccine. One capsule is swallowed on alternate days, e.g. days 30, 32, 34, and 36 for a total of 4 capsules.
  Other Names: Vivotif

SUMMARY:
The purpose of this study is to determine if adding dietary fiber, such as inulin, to a diet that does not have enough fiber would raise the levels of potentially beneficial bacteria, such as Bifidobacterium, in the gut. There is evidence to suggest that these microbes can affect gut health and immune response, including to vaccines. The investigators will examine how inulin in the diet (compared to the maltodextrin control) (1) causes changes in the composition and function of the gut microbes, (2) reduces gut inflammation and gut leakiness caused by the vaccine, (3) increases immune response to vaccination, and (4) changes the expression of important adhesion molecules on the surface of white blood cells. Intestinal and whole-body responses will be measured in all participants.

DETAILED DESCRIPTION:
Inulin, a dietary fiber supplement, is known to increase gut levels of potentially beneficial bacteria, including Bifidobacterium that are indigenous to gut microbiomes. Our underlying hypothesis is that the commensal microbiome, including Bifidobacterium, in the proximal colon or distal ileum affects the environment of draining lymph nodes and can thus modulate immune responses, including to vaccines. In the current study, participants will consume 12 grams/day inulin or maltodextrin (control) for 3 weeks before the administration of the Ty21a typhoid fever vaccine, 1 week during the vaccine, and 1 week after the vaccine. Vaccine response will be measured by counting T cells and immunoglobulin G (IgG) or immunoglobulin A (IgA)-secreting plasma cells specific for Ty21a. Gut permeability will be measured at baseline, and before and after the vaccine administration. Systemic inflammation and immune activation will be measured by analyzing blood for markers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Body Mass Index (BMI) 18.5 - 30.9 kg/m2
2. inadequate total dietary fiber intake defined as:

   * Females 18 - 30 years old, less than 28 g/day
   * Females 31 - 50 years old, less than 25 g/day
   * Females 51+ year old, less than 22 g/day
   * Males 18 - 30 years old, less than 34 g/day
   * Males 31 - 50 years old, less than 31 g/day
   * Males 51+ years old, less than 28 g/day

Exclusion Criteria:

1. blood pressure greater than or equal to 140/90 mmHg
2. has HIV/AIDS or another disease that affects the immune system
3. has any kind of cancer
4. inability to lift 30 pounds with assistance (for transporting refrigerated stool containers)
5. decline to take an HIV blood test
6. pregnant or lactating women
7. refusal to take a pregnancy test
8. female subjects: refusal to use a method of birth control 1 week prior to the administration of the vaccine, 1 week during the vaccine, and 1 week after the vaccine
9. allergy to vaccine components, i.e. thimerosal and enteric-coated capsules
10. allergy to oral typhoid vaccine
11. use of anti-inflammatory medications, i.e. nonsteroidal anti-inflammatory drugs (NSAID), aspirin, 3 or more times per month
12. use of sulfonamides or antibiotics 3 months prior to the receipt of Ty21a vaccine.
13. use of anti-hypertensive drugs, i.e. beta blockers, diuretics, calcium channel blockers
14. use of anti-malaria drugs, i.e. mefloquine, chloroquine, and proguanil
15. use of drugs that affects the immune system, i.e. immunosuppressants, immune-modifying drugs, corticosteroids, i.e. cortisone, prednisone, methylprednisolone, for 2 weeks or longer
16. use of biologics, i.e. Lantus, Remicade, Rituxan, Humira, Herceptin, Avastin, Lucentis, Enbrel for 2 weeks or longer
17. undergoing cancer treatment with radiation or drugs
18. greater than 10 years residence in a typhoid-endemic area
19. receipt of typhoid vaccine in the last 5 years
20. receipt of any vaccine two weeks prior to receipt of Ty21a vaccine
21. individuals at increased risk of developing complications from a live, bacterial vaccine
22. history of typhoid fever
23. history of primary immune deficiency or autoimmune disease
24. history of acute or chronic gastrointestinal (GI) disorder, i.e. Crohn's disease, irritable bowel syndrome, gastric ulcer
25. diarrheal illness (defined as passing 3 or more abnormally loose or watery stool in a 24 hour period) or persistent vomiting 2 weeks prior to the study
26. history of chronic illnesses, i.e. diabetes, cardiovascular disease, cancer, gastrointestinal malabsorption or inflammatory diseases, kidney disease, autoimmune disorders, HIV, liver disease, including hepatitis B and C
27. asthma if taking medication on a daily basis
28. recent surgery (within 3 months)
29. history of GI surgery
30. recent hospitalization (within 3 months)
31. fever (within 2 weeks)
32. unwillingness to discontinue probiotic, prebiotic, or other supplements (except Recommended Dietary Allowance-level vitamin and mineral supplements), fiber supplements, or food and beverage products containing inulin, chicory root fiber, or maltodextrin during the study
33. not having at least one arm vein suitable for blood drawing
34. unwilling or uncomfortable with blood draws and stool collections
35. regular blood or blood product donation and refusal to suspend donation
36. current participation in another research study
37. unable to fast for 12-16 hours
38. have fewer than 3 bowel movements per week
39. consuming one or more servings of added-inulin foods per day over the past month

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Change in vaccine-specific antibody-secreting cell response to oral Ty21a typhoid vaccination using the standard 4-dose regimen | Day 26, 37, and 39
  Measurement of baseline level (Day 26; before first vaccine dose) and post-vaccine, antibody response, Immunoglobulin G (IgG), Immunoglobulin M (IgM) and IgA, 7 and 9 days after the first vaccine dose using the antibody-in-lymphocyte-supernatant (ALS) assay to identify antibody-secreting cells in blood. Two antigens will be used: Ty21a outer membrane protein and lipopolysaccharide from Salmonella Typhi.

SECONDARY OUTCOMES:
Change in vaccine-specific serum antibody response to typhoid vaccination | Day 26 and 58
  Measurement of baseline level (Day 26; before first vaccine dose) and post-vaccine (28 d after first vaccine dose) antibody levels (IgG, IgM, IgA)
Change in vaccine-specific fecal IgA antibody levels from typhoid vaccination | Day 26, 39, and 58
  Measurement of baseline level (Day 26; before first vaccination dose) and change in fecal antibody levels
Change in plasma cytokines as markers of systemic inflammation | Day 8, 26, 37, 39, and 58
  Measurement of plasma cytokines, such as interleukin-6 (IL-6), tumor necrosis factor-alpha (TNF-alpha), and IL-1beta
Change in plasma acute phase proteins and adhesion molecules | Day 8, 26, 37, 39, and 58
  Measurement of acute phase reactants, such as C-reactive protein (CRP) and serum amyloid-A (SAA), and intercellular adhesion molecules, such as intercellular adhesion molecule-1 (ICAM-1) and vascular endothelial cell adhesion molecule-1 (VCAM-1)
Change in a plasma marker of lipopolysaccharide (LPS) exposure | Day 8, 26, 37, 39, and 58
  Measurement of plasma LPS-binding protein using an ELISA.
Change in blood monocyte subsets | Day 8, 26, 37, 39, and 58
  Monocyte subsets will be analyzed using flow cytometry.
Change in plasma short chain fatty acids (SCFA) | Day 8, 26, 37, 39, and 58
  Plasma SCFA will be measured using liquid chromatography-mass spectrometry (LC-MS).
Change in urinary lactulose and D-mannitol | Day 8, 26, and 37
  Measurement of lactulose to mannitol ratio, an indicator of intestinal permeability, in urine
Change in fecal microbiome | Period 1: Days 1-7; Period 2: Days 16-25; Period 3: Days 26-36; Period 4: Days 37-43; Period 5: Days 58-65
  Measurement of relative abundance of colonic bacteria using DNA isolated from stool.
Change in fecal mRNA | Period 1: Days 1-7; Period 2: Days 16-25; Period 3: Days 26-36; Period 4: Days 37-43; Period 5: Days 58-65
  Total RNA, and specifically, messenger ribonucleic acid (mRNA), will be analyzed from preserved stools.
Change in stool consistency and frequency | Period 1: Days 1-7; Period 2: Days 16-25; Period 3: Days 26-36; Period 4: Days 37-43; Period 5: Days 58-65
  Measurement of stool consistency using the Bristol stool scale, a medical tool used to classify stool forms into 7 categories, and frequency via self-report in diaries.
Change in GI symptoms | Period 1: Days 1-7; Period 2: Days 16-25; Period 3: Days 26-36; Period 4: Days 37-43; Period 5: Days 58-65
  Measurement of GI symptoms using a 10-symptom health questionnaire with degree of discomfort ranked in one of four categories (0 absent, 1 mild, 2 moderate, or 3 severe; PMID: 9301412)
Change in fecal pH | Period 1: Days 1-7; Period 2: Days 16-25; Period 3: Days 26-36; Period 4: Days 37-43; Period 5: Days 58-65
  Measurement of fecal pH using a standard pH meter.
Change in fecal calprotectin | Period 1: Days 1-7; Period 2: Days 16-25; Period 3: Days 26-36; Period 4: Days 37-43; Period 5: Days 58-65
  Measurement of calprotectin will be done by ELISA
Change in fecal SCFA | Period 1: Days 1-7; Period 2: Days 16-25; Period 3: Days 26-36; Period 4: Days 37-43; Period 5: Days 58-65
  Measurement of SCFA will be done by gas chromatography-mass spectrometry (GC-MS.)
Change in fecal metabolites | Period 1: Days 1-7; Period 2: Days 16-25; Period 3: Days 26-36; Period 4: Days 37-43; Period 5: Days 58-65
  Measurement of bile acids and other metabolites will be measured
Change in fecal secretory total immunoglobulin A (sIgA) | Period 1: Days 1-7; Period 2: Days 16-25; Period 3: Days 26-36; Period 4: Days 37-43; Period 5: Days 58-65
  Measurement of total fecal sIgA using ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Lemay, PhD, Principal Investigator — USDA, ARS, Western Human Nutrition Research Center; Ryan Snodgrass, PhD, Principal Investigator — USDA, ARS, Western Human Nutrition Research Center; Mary Kable, PhD, Principal Investigator — USDA, ARS, Western Human Nutrition Research Center; Bess Caswell, PhD, Principal Investigator — USDA, ARS, Western Human Nutrition Research Center
Locations (1):
- USDA, ARS, Western Human Nutrition Research Center, Davis, California, United States

REFERENCES:
- [Background] Meyer D, Stasse-Wolthuis M. The bifidogenic effect of inulin and oligofructose and its consequences for gut health. Eur J Clin Nutr. 2009 Nov;63(11):1277-89. doi: 10.1038/ejcn.2009.64. Epub 2009 Aug 19. PMID 19690573
- [Background] Costabile A, Kolida S, Klinder A, Gietl E, Bauerlein M, Frohberg C, Landschutze V, Gibson GR. A double-blind, placebo-controlled, cross-over study to establish the bifidogenic effect of a very-long-chain inulin extracted from globe artichoke (Cynara scolymus) in healthy human subjects. Br J Nutr. 2010 Oct;104(7):1007-17. doi: 10.1017/S0007114510001571. Epub 2010 Jul 1. PMID 20591206
- [Background] Dewulf EM, Cani PD, Claus SP, Fuentes S, Puylaert PG, Neyrinck AM, Bindels LB, de Vos WM, Gibson GR, Thissen JP, Delzenne NM. Insight into the prebiotic concept: lessons from an exploratory, double blind intervention study with inulin-type fructans in obese women. Gut. 2013 Aug;62(8):1112-21. doi: 10.1136/gutjnl-2012-303304. Epub 2012 Nov 7. PMID 23135760
- [Background] Holscher HD, Bauer LL, Gourineni V, Pelkman CL, Fahey GC Jr, Swanson KS. Agave Inulin Supplementation Affects the Fecal Microbiota of Healthy Adults Participating in a Randomized, Double-Blind, Placebo-Controlled, Crossover Trial. J Nutr. 2015 Sep;145(9):2025-32. doi: 10.3945/jn.115.217331. Epub 2015 Jul 22. PMID 26203099
- [Background] Kolida S, Meyer D, Gibson GR. A double-blind placebo-controlled study to establish the bifidogenic dose of inulin in healthy humans. Eur J Clin Nutr. 2007 Oct;61(10):1189-95. doi: 10.1038/sj.ejcn.1602636. Epub 2007 Jan 31. PMID 17268410
- [Background] Menne E, Guggenbuhl N, Roberfroid M. Fn-type chicory inulin hydrolysate has a prebiotic effect in humans. J Nutr. 2000 May;130(5):1197-9. doi: 10.1093/jn/130.5.1197. PMID 10801918
- [Background] Micka A, Siepelmeyer A, Holz A, Theis S, Schon C. Effect of consumption of chicory inulin on bowel function in healthy subjects with constipation: a randomized, double-blind, placebo-controlled trial. Int J Food Sci Nutr. 2017 Feb;68(1):82-89. doi: 10.1080/09637486.2016.1212819. Epub 2016 Aug 5. PMID 27492975
- [Background] Petry N, Egli I, Chassard C, Lacroix C, Hurrell R. Inulin modifies the bifidobacteria population, fecal lactate concentration, and fecal pH but does not influence iron absorption in women with low iron status. Am J Clin Nutr. 2012 Aug;96(2):325-31. doi: 10.3945/ajcn.112.035717. Epub 2012 Jun 27. PMID 22743314
- [Background] Huda MN, Lewis Z, Kalanetra KM, Rashid M, Ahmad SM, Raqib R, Qadri F, Underwood MA, Mills DA, Stephensen CB. Stool microbiota and vaccine responses of infants. Pediatrics. 2014 Aug;134(2):e362-72. doi: 10.1542/peds.2013-3937. Epub 2014 Jul 7. PMID 25002669
- [Background] Huda MN, Ahmad SM, Alam MJ, Khanam A, Kalanetra KM, Taft DH, Raqib R, Underwood MA, Mills DA, Stephensen CB. Bifidobacterium Abundance in Early Infancy and Vaccine Response at 2 Years of Age. Pediatrics. 2019 Feb;143(2):e20181489. doi: 10.1542/peds.2018-1489. PMID 30674610
- [Background] Zuckerman JN, Hatz C, Kantele A. Review of current typhoid fever vaccines, cross-protection against paratyphoid fever, and the European guidelines. Expert Rev Vaccines. 2017 Oct;16(10):1029-1043. doi: 10.1080/14760584.2017.1374861. PMID 28856924
- [Background] Fiorentino M, Lammers KM, Levine MM, Sztein MB, Fasano A. In vitro Intestinal Mucosal Epithelial Responses to Wild-Type Salmonella Typhi and Attenuated Typhoid Vaccines. Front Immunol. 2013 Feb 12;4:17. doi: 10.3389/fimmu.2013.00017. eCollection 2013. PMID 23408152
- [Background] Salerno-Goncalves R, Galen JE, Levine MM, Fasano A, Sztein MB. Manipulation of Salmonella Typhi Gene Expression Impacts Innate Cell Responses in the Human Intestinal Mucosa. Front Immunol. 2018 Nov 1;9:2543. doi: 10.3389/fimmu.2018.02543. eCollection 2018. PMID 30443257

DOCUMENTS (1):
  • Informed Consent Form (2025-03-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT04543877/ICF_000.pdf